CLINICAL TRIAL: NCT06909604
Title: Al18F-HER2-BCH PET/CT to Predict Response in Breast Patients Treated With Neoadjuvant Therapy
Brief Title: Al18F-HER2-BCH PET in Breast Patients Treated With Neoadjuvant Therapy
Acronym: HERfore
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: The Affiliated Hospital of Qingdao University (Other); North Sichuan Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2019KT114-ZY02
Record Dates: First submitted 2024-12-24; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: breast cancer; PET/CT; Neoadjuvant therapy; HER2 expression
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HER2 expression of PET imaging (Experimental): Evaluate the diagnostic potential of HER2 imaging using 18F-labelled HER2 affibody , evaluate the predictive and prognostic value of HER2 PET imaging in breast cancer patients treated with neoadjuvant therapy
  Interventions: Radiation: HER2 expression of PET imaging

INTERVENTIONS:
Radiation: HER2 expression of PET imaging — Evaluate the diagnostic potential of HER2 imaging using 18F-labelled HER2 affibody , evaluate the predictive and prognostic value of HER2 PET imaging in bladder cancer patients treated with neoadjuvant therapy

SUMMARY:
To use the molecular PET radionuclide (F-18) labelled HER2 Affibody to evaluate the predictive and prognostic value in breast patients treated with neoadjuvant therapy

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years old; ECOG 0 or 1;
2. Patients with newly diagnosis HER2 positive or suspicious positive tumors;
3. Receives neoadjuvant therapy
4. Has adequate cardiac, bone marrow, renal, hepatic and blood clotting functions;
5. Life expectancy > 3 months -

Exclusion Criteria:

1. Significant hepatic or renal dysfunction;
2. Is pregnant or ready to pregnant;
3. Cannot keep their states for half an hour;
4. Refused to join the clinical research;
5. Suffering from claustrophobia or other mental disorders;
6. Any other situation that researchers considered it unsuitable to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in SUVmax before and after treatment | Before treatment, 9 weeks after treatment, before surgery
  The uptake of the tracer in the primary and metastatic tumor lesions by measuring standardized uptake value (SUV) on PET/CT

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, China